CLINICAL TRIAL: NCT02094963
Title: A Randomized, Open-label, Parallel Group, Multicenter Phase IV Study to Assess Safety and Efficacy of Ticagrelor Versus Clopidogrel in Asian/KOREAn Patients With Acute Coronary Syndromes Intended for Invasive Management:TICAKOREA Trial
Brief Title: Safety and Efficacy of Ticagrelor Versus Clopidogrel in Asian/KOREAn Patients With Acute Coronary Syndromes Intended for Invasive Management
Acronym: TICA KOREA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, MD, PhD, Asan Medical Center
Organization: Asan Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMCCV2013-14
Record Dates: First submitted 2014-03-10; First posted 2014-03-24 (Estimated); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Acute Coronary Syndrome; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Angina Pectoris
Keywords: acute coronary syndrome; coronary disease; coronary artery disease
MeSH Terms: conditions — Acute Coronary Syndrome; Myocardial Ischemia; Heart Diseases; Cardiovascular Diseases; Angina Pectoris; Coronary Disease; Coronary Artery Disease | interventions — Ticagrelor; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ticagrelor (Experimental)
  Interventions: Drug: Ticagrelor
- Clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Ticagrelor — 180mg loading and 90mg bid
  Arms: Ticagrelor
Drug: Clopidogrel — 600mg loading and 75mg qd
  Arms: Clopidogrel

SUMMARY:
The purpose of this study is to assess safety and efficacy of Ticagrelor versus Clopidogrel in Asian/KOREAn patients with acute coronary syndromes intended for invasive management.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and more
* Index event of non-ST or ST segment elevation ACS
* Provision of signed informed consent

Exclusion Criteria:

* Hypersensitivity to aspirin or ticagrelor
* Oral anticoagulation therapy that cannot be stopped
* Treated with thrombolysis within 24hrs
* Any other reason the investigator deems the subject to be unsuitable for the study e.g., Active malignant tumor
* Concomitant therapy with strong CYP3A inhibitors, CYP3A substrates with narrow therapeutic index, or strong CYP3A inducers
* Any life-threatening condition with life expectancy less than 6months
* Mental condition (dementia, alcohol or drug abuse) which may be affect study compliance or prevent understanding of the aims, investigational procedures or possible consequences of the study
* High risk due to malignant hypertension
* The conditions associated with increased risk of bradycardiac events
* Subjects with severe liver disease
* Subjects requiring dialysis
* Increased bleeding risk
* History of cerebral hemorrhage, gastrointestinal bleeding within 6months, major surgical procedure within 30days
* Thrombocytopenia or leukopenia
* Positive pregnancy test or is known to be pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Actual)
Dates: Start 2014-07-05 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
The time to first occurrence of any bleeding event | 1year
  Safety of Ticagrelor compared to Clopidogrel by measuring the time to first occurrence of any bleeding event(including major, minor bleedings)
The time to first occurrence of any event from the composite of death from vascular causes, Myocardial Infarction (MI) and stroke | 1year
  Effect of Ticagrelor compared to Clopidogrel by measuring: time to first occurrence of any event from the composite of death from vascular causes, Myocardial Infarction (MI) and stroke

SECONDARY OUTCOMES:
The time to first occurrence of major bleeding event | 1year
  by PLAtelet inhibition and patient Outcomes(PLATO) criteria
The time to first occurrence of minor bleeding event | 1year
  by PLAtelet inhibition and patient Outcomes(PLATO) criteria
The time to first occurrence of major bleeding event or minor bleeding event | 1year
  The Thrombolysis in Myocardial Infarction (TIMI) bleeding criteria
The time to first occurrence of major bleeding event | 1year
  The Thrombolysis in Myocardial Infarction (TIMI) bleeding criteria
The time to first occurrence of minor bleeding event | 1year
  The Thrombolysis in Myocardial Infarction (TIMI) bleeding criteria
The time to first occurrence of Bleeding Academic Research Consortium (BARC) bleeding event from type 1 to type 5 | 1year
  By Bleeding Academic Research Consortium(BARC) Definition of Bleeding Events
The time of first occurrence of discontinuation of study medication from any bleeding event | 1year
Non serious adverse events | 1year
Adverse events following discontinuation of study medication | 1year
Serious adverse events | 1year
The time to first occurrence of death from vascular causes | 1year
  Effect of Ticagrelor compared to Clopidogrel by measuring: time to first occurrence of death from vascular causes
The time to first occurrence of myocardial infarction | 1year
  Effect of Ticagrelor compared to Clopidogrel by measuring: time to first occurrence of myocardial infarction
The time to first occurrence of stroke | 1year
  Effect of Ticagrelor compared to Clopidogrel by measuring: time to first occurrence of stroke
The time to occurrence of composite events | 1year
  The time to occurrence of composite events(death from any cause, myocardial infarction, stroke)
The time to occurrence of death from any cause | 1year
Number of patients with net clinical benefit of any total bleeding and any event from the composite of death from vascular causes, Myocardial Infarction and stroke. | 1year

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - Asan Medical Center, Seoul, Songpa-gu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Dongguk University Gyeongju Hospital, Gyeongju
  - Inje University Ilsan Paik Hospital, Ilsan
  - Gachon University Gil Hospital, Incheon
  - ChonBuk National University Hospital, Jeonju
  - Dong-A Medical Center, Pusan
  - Inje University Pusan Paik Hospital, Pusan
  - Ulsan University Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No
This is not a publicly funded trial.

REFERENCES:
- [Derived] Jang MH, Kim AR, Kim T, Oh HJ, Lee JH, Lee YJ, Kim S, Lee J, Kim JH, Cha SJ, Kim TO, Kang DY, Lee PH, Ahn JM, Park DW, Park SJ; TICAKOREA Investigators. Age- and Sex-Specific Disparities in Outcomes After Ticagrelor Versus Clopidogrel in East Asian Patients. Am J Cardiol. 2023 Nov 15;207:237-244. doi: 10.1016/j.amjcard.2023.08.124. Epub 2023 Sep 26. PMID 37757520
- [Derived] Lee J, Kim MJ, Kim M, Park J, Kim H, Cho S, Choi Y, Lee J, Kim JH, Cha SJ, Kim TO, Kang DY, Lee PH, Ahn JM, Park SJ, Park DW; TICAKOREA Study Investigators. Validation of Academic Research Consortium for High Bleeding Risk Definition in East-Asian Patients. JACC Asia. 2023 Feb 7;3(3):390-399. doi: 10.1016/j.jacasi.2022.11.012. eCollection 2023 Jun. PMID 37323862
- [Derived] Choi Y, Kang DY, Lee J, Lee J, Kim M, Kim H, Park J, Cho S, Lee J, Cha SJ, Kim TO, Lee PH, Ahn JM, Park SJ, Park DW; TICA KOREA Investigators. Ticagrelor Versus Clopidogrel in East Asian Patients With Acute Coronary Syndrome and Diabetes Mellitus. JACC Asia. 2022 Nov 15;2(6):666-674. doi: 10.1016/j.jacasi.2022.07.005. eCollection 2022 Nov. PMID 36444315
- [Derived] Park DW, Kwon O, Jang JS, Yun SC, Park H, Kang DY, Ahn JM, Lee PH, Lee SW, Park SW, Choi SW, Lee SG, Yoon HJ, Ahn T, Kim MH, Nah DY, Lee SY, Chae JK, Park SJ; TICAKOREA Investigators. Clinically Significant Bleeding With Ticagrelor Versus Clopidogrel in Korean Patients With Acute Coronary Syndromes Intended for Invasive Management: A Randomized Clinical Trial. Circulation. 2019 Dec 3;140(23):1865-1877. doi: 10.1161/CIRCULATIONAHA.119.041766. Epub 2019 Sep 25. PMID 31553203